CLINICAL TRIAL: NCT04458870
Title: Internet-based Acceptance and Commitment Therapy for Family Caregivers of People With Dementia
Brief Title: Acceptance and Commitment Therapy for Family Caregivers of People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Areum Han, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300005230
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Psychological Distress
Keywords: Caregivers; Dementia; Alzheimer's Disease; Burden; Quality of life; Acceptance and Commitment Therapy; Mindfulness; Psychological health
MeSH Terms: conditions — Dementia; Alzheimer Disease; Psychological Well-Being | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acceptance and Commitment Therapy (Experimental)
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Participants will receive 10 weekly individual acceptance and commitment therapy by a trained coach through zoom video-conferencing.

SUMMARY:
The pilot project aims to investigate the feasibility and the preliminary efficacy of a guided online acceptance and commitment therapy (ACT) intervention for distressed family caregivers of people with dementia. A one-group pretest-posttest design (n=15) will be used to investigate the potential effects of the 10 weekly online ACT intervention session on caregivers' outcomes at posttest (10 weeks).

DETAILED DESCRIPTION:
This project will employ one-group pretest-posttest design to investigate the potential impact of a guided online ACT intervention on improving quality of life and psychological health in distressed family caregivers of people with dementia. After the baseline evaluation, eligible caregivers will receive 10 weekly ACT sessions, individually delivered by a licensed professional counselor online. Each session lasts for one hour. Primary outcome measures will be psychological distress measured by the Depression, Anxiety and Stress Scale (DASS)- 21 and care-related quality of life measured by the Care-related Quality of Life instrument (CarerQol). A one-time interview at the completion of the 10 weekly sessions will be conducted to explore caregivers' experiences in the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. community-dwelling adults (age 18 or over) who are currently taking primary responsibility for the care of a relative with dementia living in the community
2. devoting at least 1 hour daily to the care of the relative with dementia
3. having cared for a relative with dementia for at least 3 months
4. suffering at least mild symptoms of psychological distress measured by the DASS-21 (scores ≥ 5 on Depression Subscale of DASS-21, scores ≥ 4 on Anxiety Subscale, or scores ≥ 8 on Stress Subscale)
5. having a computer/smartphone with internet access capable of doing web browsing and video-conferencing
6. being able to provide informed consent by understanding the nature of study participation.

Exclusion Criteria:

1. having cognitive, physical, or sensory deficits, or language barriers (non-English communicator) that impede study participation
2. receiving a psychological therapy currently
3. having psychiatric hospitalizations or diagnoses of mental illness in the previous 2 years
4. taking antipsychotic or anticonvulsant medication at the time of recruitment
5. considering or planning to place family members of dementia in a nursing home within 6 months
6. having the possibility of study dropouts due to other medical conditions of family members with dementia (e.g., conditions that may impede study participation due to frequent hospitalization or death).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
Depression, Anxiety and Stress Scale - 21 | Change from baseline to 10 weeks
  The Depression, Anxiety and Stress Scale (DASS)- 21 is a 21-item self report instrument designed to measure the three related negative emotional states of depression, anxiety and stress. Higher scores represent greater symptomatology.
Care-related Quality of Life instrument | Change from baseline to 10 weeks
  Care-related Quality of Life instrument (CarerQol) assesses the impact of providing informal care on caregivers and combines a 7-item subjective burden measure (CarerQol-7D) with well-being (CarerQol-VAS). Higher scores indicate higher levels of quality of life.

SECONDARY OUTCOMES:
Zarit Burden Interview | Change from baseline to 10 weeks
  The Zarit Burden Interview (ZBI) is a 12-item self-report questionnaire assessing caregiver. Higher scores indicate higher levels of burden.
Brief Coping Orientation to Problems Experienced | Change from baseline to 10 weeks
  Brief COPE (Coping Orientation to Problems Experienced) is a 28-item self-report questionnaire measuring coping strategies in response to stressors. Three composite subscales include problem-focused, emotion-focused, and dysfunctional coping strategies. Higher scores on a subscale indicates more frequent use of the relevant coping strategies.
Engagement in Meaningful Activities Survey | Change from baseline to 10 weeks
  The Engagement in Meaningful Activities Survey (EMAS) is a 12-item self-assessment instrument that measures a person's subjective experience of the meaningfulness of everyday activities. Higher scores indicate greater levels of engagement in meaningful activities.
Experiential Avoidance in Caregiving Questionnaire | Change from baseline to 10 weeks
  The Experiential Avoidance in Caregiving Questionnaire (EACQ) is a 15-item self-report questionnaire measuring experiential avoidance in caregivers. Higher scores indicate greater levels of experiential avoidance.
Acceptance and Action Questionnaire-II | Change from baseline to 10 weeks
  The Action and Acceptance Questionnaire (AAQ)-II is a 7-item self-report questionnaire measuring psychological flexibility. Higher scores indicate poor psychological flexibility.
Cognitive Fusion Questionnaire | Change from baseline to 10 weeks
  The Cognitive Fusion Questionnaire (CFQ)-7 is a 7-item self-report questionnaire measuring cognitive fusion. Higher scores indicate greater levels of cognitive fusion.

OTHER OUTCOMES:
Cortisol levels by collecting fingernails | Change from baseline to 10 weeks
  A biological measure of stress will be assessed through analysis of cortisol levels in caregivers' nail samples.
System Usability Scale | at 10 weeks
  The System Usability Scale (SUS) is a 10-item self-report questionnaire measuring usability of a program/intervention. Higher scores indicate greater levels of perceived usability of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Areum Han, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No